CLINICAL TRIAL: NCT06000813
Title: REACH-Es: Adapting a Digital Health Tool to Improve Diabetes Medication Adherence Among Latino Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jacqueline A. Seiglie, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023p001968; 1K23DK135798-01 (NIH)
Record Dates: First submitted 2023-08-04; First posted 2023-08-21 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Type 2 Diabetes (Adult Onset); Medication Adherence
Keywords: Type 2 diabetes; Medication adherence; Mobile health; Latino adults
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- REACH-Es (Experimental): Participants in the REACH-Es arm will receive REACH-Es short message service (SMS), as follows: 1) Daily SMS (information related to diet, exercise, self-monitoring of blood glucose, their specific diabetes medication(s), and top 4 medication adherence barriers); 2) Daily two-way SMS (diabetes medication adherence question); 3) Weekly one-way SMS (participants receive weekly feedback on Sunday regarding how many of the last 7 days they took their medicine); 4) A SMS each time an HbA1c is collected with a link to a secure website that displays the result.
  Interventions: Behavioral: REACH-Es
- Enhanced treatment as usual (ETAU) (Active Comparator): Participants will maintain care as usual (medication treatment and physician monitoring) in addition to a welcome SMS following enrollment, a SMS each time an HbA1c is collected with a link to a secure website that displays the result, and bi-monthly information on diabetes self-care education.
  Interventions: Behavioral: ETAU

INTERVENTIONS:
Behavioral: REACH-Es — REACH-Español is a mobile health platform adapted from the original REACH intervention to a Latino population with type 2 diabetes. The goal of REACH-Español is to improve diabetes medication adherence and glycemic management in this population.
  Other Names: REACH-Español
  Arms: REACH-Es
Behavioral: ETAU — Participants will maintain care as usual (medication treatment and physician monitoring) in addition to a welcome SMS following enrollment, a SMS each time an HbA1c is collected with a link to a secure website that displays the result, and bi-monthly information on diabetes self-care education.
  Arms: Enhanced treatment as usual (ETAU)

SUMMARY:
Latino individuals, the fastest growing ethnic minority population in the United States, have a higher prevalence of type 2 diabetes and diabetes-related complications, and are more likely to report inconsistent use of diabetes medications than non-Hispanic White individuals. The proposed project will test an interactive text message-based tool tailored to address barriers to taking diabetes medications that are relevant to Latino adults. If found feasible, acceptable, and usable, this intervention could serve as a scalable tool to improve diabetes management and reduce diabetes-related complications among Latino adults in the United States.

DETAILED DESCRIPTION:
Latino adults have a disproportionate burden of type 2 diabetes and diabetes-related complications. Diabetes medication non-adherence is an important modifiable contributor to suboptimal glycemic management among Latino adults, who are nearly twice as likely to report non-adherence to diabetes medications as non-Hispanic White individuals. Besides language barriers, additional commonly reported barriers that contribute to non-adherence in this population include negative perceptions about insulin use and misunderstanding ongoing need for diabetes medications once HbA1c has improved. Mobile health (mHealth) technology can reduce medication adherence barriers and improve adherence behavior, but mHealth tools that address commonly reported barriers to diabetes medication adherence among Latino adults are lacking. One such mHealth platform is REACH (Rapid Encouragement/Education And Communications for Health), a text message-based tool that improved diabetes medication adherence and glycemic control among English-speaking adults with type 2 diabetes.

This study will evaluate REACH-Español (hereafter "REACH-Es), an mHealth platform adapted from the original REACH intervention that will incorporate qualitative input from Latino adults with type 2 diabetes on barriers to diabetes medication adherence relevant to this population. Specifically, the investigators will conduct a pilot RCT (n=70) to assess feasibility, acceptability, and usability of REACH-Es, as well as intervention targets (diabetes medication adherence and barriers to adherence) comparing REACH-Es to enhanced treatment as usual; secondary outcomes are HbA1c and diabetes self- efficacy. The project will generate preliminary data for an R01 hybrid-effectiveness implementation trial of REACH-Es.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Have current or prior (since 2018) HbA1c ≥8.0%
* Take at least one diabetes medication
* Receive care at MGH- affiliated primary care practices (≥2 visits in the past 3 years)
* ≥18 yrs
* Identify as Latino and/or Hispanic
* Speak and read in Spanish as preferred language
* Willing and able to provide informed consent
* Access to a mobile telephone with text messaging capability
* Suboptimal diabetes medication adherence, assessed using the first 2 items in the Adherence to Refill and Medication Scale (ARMS-d) questionnaire combined: "How frequently do you forget or decide to not take your diabetes medications?" Participants who answer sometimes, almost always, and/or always will be considered eligible for the study.

Exclusion Criteria:

* Auditory limitations and/or inability to communicate orally
* Inability to receive, read, or send a text message (assessed by a trained research assistant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Feasibility (recruitment rate) | Collected at 0 months
  Number of eligible participants who enroll/ Number of eligible participants who are contacted and reached by phone
Feasibility (response rate to 2-way text messages) | Collected at 3 and 6 months
  Number of 2-way text messages answered/ Number of 2-way text messages received
Feasibility (retention rate) | Collected at 3 and 6 months
  Number of participants enrolled in the study at follow-up/ Number of participants enrolled at the start of the study
Acceptability | Collected at 3 and 6 months
  Assessed quantitatively based on utility of REACH-Es on a 0-10 Likert scale and qualitatively through exit interviews.
Usability | Collected at 3 and 6 months
  Assessed quantitatively by administering the 10-item Spanish version of the System Usability Scale (SUS) questionnaire, scored on a 0-5 Likert-type scale.
Diabetes Medication adherence | Collected at 0, 3, and 6 months
  Assessed using the 11-item Adherence to Refill and Medication Scale (ARMS-d) questionnaire scored on a 0-4 Likert scale (range 12-48).
IMB barrier sum score | Collected at 0, 3, and 6 months
  Calculated by rating each barrier item on a 0-10 scale (1=never to 10=a lot) and identifying each participant's 4 highest- scored barriers (range 4-40).

SECONDARY OUTCOMES:
HbA1c | Collected at 0, 3, and 6 months
  The HbA1c collection will be done through: 1) EHR review if available <3 weeks from the enrollment visit, 2) point-of-care testing; or) clinical lab draw.
Diabetes self-efficacy | Collected at 0, 3, and 6 months
  Assessed by administering the 8-item Spanish Diabetes Self-Efficacy questionnaire (0-10 Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Seiglie, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Diabetes Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD can be requested by qualified investigators with interest in type 2 diabetes. Access to the data will be contingent on review and approval of a research proposal and Statistical Analysis Plan.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be made 12 months after manuscript publication and will be made available for up to 24 months.
Access Criteria: Access to the data will be contingent on review and approval of a research proposal and Statistical Analysis Plan.